CLINICAL TRIAL: NCT05500859
Title: Swiss Secondary Prevention and Rehabilitation Registry: SwissPR
Brief Title: Swiss Secondary Prevention and Rehabilitation Registry
Acronym: SwissPR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02057; me19Pfister
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases (CVD)
Keywords: Coronary artery disease (CAD); Cardiac rehabilitation (CR); Acute coronary syndrome (ACS); Chronic coronary syndrome (CCS); Prevention benchmark performance measures (BPM); KARAMBA; Swiss Prevention and Rehabilitation Registry (SwissPR)
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Acute Coronary Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection at Baseline, 3 months after baseline (BL), 1-year follow-up, Telephone follow-up and questionnaire 3 years and 5 years after BL — Data collection (Patient characteristics including medical history, current medication, cardiovascular risk factors, routine laboratory analysis (including lipids, Hb1c, NT-proBNP), clinical status, electrocardiogram, echocardiography data from latest echo, cardio pulmonary exercise testing (CPET), questions on general health behavior (diet, weekly exercise load), Quality of Life and questions on socio-economic parameters)

SUMMARY:
The SwissPR study is to continuously monitor patient characteristics and short- and long-term benchmark quality measures and outcomes of patients participating in a 12-week ambulatory CR program.

DETAILED DESCRIPTION:
The SwissPR study is a non-interventional, longitudinal observational cohort study consisting of a retrospective and a prospective part of patients who have completed the Cardiac Rehabilitation (CR) program of the University Hospital Basel. Assessing the impact of a CR program on key cardiovascular Benchmark Performance Measures (BPM) and its persistence over time would be helpful on internal quality control as well as identification of special need patients with highest cardiovascular risk. "KARAMBA" is the outpatient cardiovascular prevention and rehabilitation program of the University Hospital Basel (USB) and is one of the largest CR centers in Switzerland. Data regarding the Swiss population during and after CR is missing so far, thus creating a Swiss Prevention and Rehabilitation Registry (= SwissPR) on the basis of the KARAMBA infrastructure has the potential to collect missing data and address these questions. The results of the study will identify patient profiles at increased risk (special need patients) and will shed light into the mechanisms of poor secondary prevention behavior. The objective of SwissPR is to continuously monitor patient characteristics and short- and long-term benchmark quality measures and outcomes of patients participating in a 12-week ambulatory CR program.

For the prospective and retrospective part no recruitment or screening procedure is required. The procedure of enrolling patients for the prospective cohort of SwissPR patients is based on the participation in the CR program of the University Hospital Basel. Patients are routinely referred by various institutions for participation in the CR program according to predefined cardiovascular diagnosis. The retrospective part applies to data of patients, which have completed the CR program in Basel between 2017 and 2019.

Procedures:

Visit 1: Baseline, start of ambulatory CR program (approx. 60min): Patient characteristics including medical history, current medication, cardiovascular risk factors, routine laboratory analysis (including lipids, Hb1c, NT-proBNP), clinical status, electrocardiogram, echocardiography data from latest echo, cardio pulmonary exercise testing (CPET), questions on general health behavior (diet, weekly exercise load), Quality of Life and questions on socio-economic parameters.

Visit 2: End of CR program, 3 months after baseline (approx. 60 min.): Same measurements and procedures as at visit 1.

Visit 3: 1-year follow-up (approx. 15 min.): Same measurements and procedures as at visit 1 and 2 except for CPET.

Telephone follow-up and questionnaire 3 years after CR (approx. 15 min.): After checking vital status, the following end-points and information will be collected by telephone interview: hospitalisations since last follow-up (cardiac, non-cardiac), Major Cardiovascular Adverse Events (MACE) including cardiovascular mortality, myocardial infarction, stroke, revascularization, hospitalization for heart failure, smoking status and physical activity. The questionnaire contains questions on health behaviour, quality of life, depression and medication.

Telephone follow-up and questionnaire 5 years after CR (approx. 15 min.): Same interview and questionnaire as at 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participation in an ambulatory CR program (all age groups)
* Written informed consent

Exclusion Criteria:

* Inability to follow an ambulatory CR program more than 3 weeks
* Not willing to give informed consent
* Inability to understand the informed consent due to language comprehension
* Lack of discernment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The procedure of enrolling patients for the prospective cohort of SwissPR patients is based on the participation in the CR program of the University Hospital Basel. Patients are routinely referred by various institutions for participation in the CR program according to predefined cardiovascular diagnosis.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Change in Guideline recommended medical therapy | 1 year
  Change in Guideline recommended medical therapy (Guideline recommended medical therapy is one variable in predefined secondary prevention benchmark performance measures (BPM) at one year after CR)
Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: LDL-Cholesterol target value | 1 year
  Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: LDL-Cholesterol target value
Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: blood-pressure (systolic and diastolic) | 1 year
  Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: Achievement of target blood-pressure
Change in smoking status | 1 year
  Change in smoking status (smoking status is a predefined secondary prevention benchmark performance measures (BPM) at one year after CR: Achievement of Non-smoking status)
Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: exercise/ week | 1 year
  Change in predefined secondary prevention benchmark performance measures (BPM) at one year after CR: Achievement of 150 minutes of exercise/ week (self-reported)

SECONDARY OUTCOMES:
Percentage of patients reaching the predefined secondary prevention benchmark after CR | 3 months after baseline
  Percentage of patients reaching the predefined secondary prevention benchmark after CR
Change in physical activity | up to 5 years
  Change in physical activity (measured by exercise capacity (Watt) since last follow-up
Change in medical therapy between visits | up to 5 years
  Change in medical therapy between visits
Change in quality of life questionnaire/ score between visits | up to 5 years
  Change in quality of life questionnaire between visits. The questionnaire covers various attributes of an individuals life, summing the items for each life area for a total score (possible score range 0-96).
Change in Thrombolysis in Myocardial Infarction Risk Score for Secondary Prevention (TRS 2P) between visits | up to 5 years
  Change in Thrombolysis in Myocardial Infarction Risk Score for Secondary Prevention (TRS 2P): 3 categories: G1 (Low-risk; TRS-2P = 0/1); G2 (Intermediate-risk; TRS-2P = 2); and, G3 (High-risk; TRS-2P ≥ 3)
Change in total mortality after 1, 3 and 5 years | up to 5 years
  Number of total mortality after 1, 3 and 5 years
Change in total MACE after 1, 3 and 5 years | up to 5 years
  Change in total MACE after 1, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Otmar Pfister, Prof. Dr. med., Principal Investigator — Outpatient Cardiology, University Hospital Basel
Locations (1):
- University Hospital Basel, Division of Outpatient Cardiology, Basel, Switzerland